CLINICAL TRIAL: NCT03272347
Title: A Phase 2B, Randomized, Double-Blind, Active-Comparator-Controlled, Dose-Ranging Clinical Trial to Evaluate the Safety, Tolerability, Antiretroviral Activity, and Pharmacokinetics of MK-8591 Given in Combination With Doravirine (DOR) and Lamivudine (3TC) in HIV-1-Infected Treatment-Naïve Adults
Brief Title: Islatravir (MK-8591) With Doravirine and Lamivudine in Participants Infected With Human Immunodeficiency Virus Type 1 (MK-8591-011)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591-011; 2017-000437-32 (EudraCT Number)
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — islatravir; doravirine; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking in Part 1, including matching placebo. Masking only to dose in Part 2. No masking in Parts 3 and 4.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Islatravir 0.25 mg (Experimental): Participants will be treated once daily (QD) with 0.25 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to doravirine/lamivudine/tenofovir disoproxil fumarate (DOR/3TC/TDF) for a minimum of 24 weeks. Between week 24 through week 52, 3TC and placebo to DOR/3TC/TDF may be discontinued. Around Week 60, participants may be switched to a selected open label dose of islatravir and DOR 100 mg QD and continue treatment until Week 144. At Week 144 participants will receive the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label and will continue treatment until Week 192.
  Interventions: Drug: Islatravir; Drug: Doravirine; Drug: Lamivudine; Drug: Placebo to Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate; Drug: Doravirine/Islatravir
- Islatravir 0.75 mg (Experimental): Participants will be treated QD with 0.75 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. Between week 24 through week 52, 3TC and placebo to DOR/3TC/TDF may be discontinued. Around Week 60, participants may be switched to a selected open label dose of islatravir and DOR 100 mg QD and will continue treatment until Week 144. At Week 144 participants will receive the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label and will continue treatment until Week 192.
  Interventions: Drug: Islatravir; Drug: Doravirine; Drug: Lamivudine; Drug: Placebo to Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate; Drug: Doravirine/Islatravir
- Islatravir 2.25 mg (Experimental): Participants will be treated QD with 2.25 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. Between week 24 through week 52, 3TC and placebo to DOR/3TC/TDF may be discontinued. Around Week 60, participants may be switched to a selected open label dose of islatravir and DOR 100 mg QD and will continue treatment until Week 144. At Week 144 participants will receive the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label and will continue treatment until Week 192.
  Interventions: Drug: Islatravir; Drug: Doravirine; Drug: Lamivudine; Drug: Placebo to Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate; Drug: Doravirine/Islatravir
- DOR/3TC/TDF (Active Comparator): Participants will be treated QD with placebo to islatravir, placebo to DOR, placebo to 3TC, and a fixed dose combination of DOR/3TC/TDF consisting of 100 mg DOR + 300 mg 3TC + 300 mg TDF for a minimum of 24 weeks. Between week 24 through week 52 placebo treatments may be discontinued and participants will receive only DOR/3TC/TDF QD open label up to Week 144. At Week 144 participants will receive the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label and will continue treatment until Week 192.
  Interventions: Drug: Placebo to Islatravir; Drug: Placebo to Doravirine; Drug: Placebo to Lamivudine; Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate; Drug: Doravirine/Islatravir

INTERVENTIONS:
Drug: Islatravir — Islatravir at 0.25 mg, 0.75 mg or 2.25 mg is orally administered QD in capsule form for up to 52 weeks. After Week 60 a selected open label dose may be administered.
  Other Names: MK-8591
  Arms: Islatravir 0.25 mg; Islatravir 0.75 mg; Islatravir 2.25 mg
Drug: Placebo to Islatravir — Placebo to islatravir is orally administered QD in capsule form for up to 52 weeks
  Arms: DOR/3TC/TDF
Drug: Doravirine — Doravirine 100 mg is orally administered QD in tablet form for up to 144 weeks
  Other Names: MK-1439
  Arms: Islatravir 0.25 mg; Islatravir 0.75 mg; Islatravir 2.25 mg
Drug: Placebo to Doravirine — Placebo to Doravirine is orally administered QD in tablet form for up to 52 weeks
  Arms: DOR/3TC/TDF
Drug: Lamivudine — Lamivudine 300 mg is orally administered QD in tablet form for up to 52 weeks
  Other Names: 3TC
  Arms: Islatravir 0.25 mg; Islatravir 0.75 mg; Islatravir 2.25 mg
Drug: Placebo to Lamivudine — Placebo to Lamivudine is orally administered QD in tablet form for up to 52 weeks
  Arms: DOR/3TC/TDF
Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate — Fixed dose combination of 100 mg doravirine + 300 mg lamivudine + 300 mg tenofovir disoproxil fumarate is orally administered QD in tablet form for up to 144 weeks.
  Other Names: MK-1439A
  Arms: DOR/3TC/TDF
Drug: Placebo to Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate — Placebo to doravirine/lamivudine/tenofovir disoproxil fumarate is orally administered QD in tablet form for up to 52 weeks
  Arms: Islatravir 0.25 mg; Islatravir 0.75 mg; Islatravir 2.25 mg
Drug: Doravirine/Islatravir — Fixed dose combination of islatravir 0.75 mg/doravirine 100 mg orally administered QD in tablet form for 48 weeks
  Other Names: MK-8591A

SUMMARY:
This study will evaluate the safety, tolerability, antiretroviral activity, and pharmacokinetics of 3 doses of islatravir (MK-8591) in combination with doravirine (DOR) and lamivudine (3TC) administered to antiretroviral treatment-naïve adult participants with human immunodeficiency virus type 1 (HIV-1) infection.

ELIGIBILITY:
Inclusion Criteria:

* Has HIV-1 infection
* Is naïve to anti-retroviral therapy (ART).
* Is clinically stable, with no signs or symptoms of acute infection, at the time of entry into the study
* Female is not pregnant, not breastfeeding, not a woman of childbearing potential (WOCBP); but if WOCBP agrees to follow the contraceptive guidance
* All participants, male and female, agree to use barrier methods of contraception when engaged in any sexual activity during treatment and for 6 weeks following treatment.

Exclusion Criteria:

* Is a user of recreational or illicit drugs or has had a history of drug or alcohol abuse or dependence that may interfere with trial participation
* Has significant hypersensitivity or other contraindication to any of the components of the study drugs
* Has a history of malignancy ≤5 years prior
* Female expects to donate eggs at any time during the study
* Is breastfeeding or expecting to conceive
* A WOCBP who has a positive urine pregnancy test on Day 1 before the first dose of study treatment
* Has been treated for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1
* Has used systemic immunosuppressive therapy or immune modulators within 30 days prior to treatment in this study or is anticipated to need them during the course of the study
* Requires any of the following prohibited medications: Carbamazepine, Phenobarbital, Phenytoin, Rifabutin, Rifampin, Herbal remedies, St. John's Wort, Modafinil, Bosentan, Nafcillin, Pentostatin
* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days of signing informed consent to participate in this current trial
* Has a documented or known virologic resistance to any approved HIV-1 reverse transcriptase inhibitor, protease inhibitor, integrase inhibitor
* Has active hepatitis C virus (HCV) coinfection defined as detectable HCV RNA or HBV co-infection defined as hepatitis B surface antigen [HBsAg]-positive
* Has a current (active) diagnosis of acute hepatitis due to any cause
* Has previously been randomized in a study and received islatravir (MK-8591), DOR, Doravirine, Tenofovir, Lamivudine, or 3TC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (26):
- United States (10):
  - Pueblo Family Physicians ( Site 0119), Phoenix, Arizona
  - University California / Davis ( Site 0101), Sacramento, California
  - Whitman Walker Clinic ( Site 0108), Washington D.C., District of Columbia
  - Orlando Immunology Center (OIC) ( Site 0105), Orlando, Florida
  - Northstar Medical Center ( Site 0102), Chicago, Illinois
  - Kansas City CARE Clinic ( Site 0106), Kansas City, Missouri
  - Saint Hope Foundation, Inc. ( Site 0116), Bellaire, Texas
  - North Texas Infectious Diseases Consultants, PA ( Site 0103), Dallas, Texas
  - Tarrant County Infectious Disease Associates ( Site 0112), Fort Worth, Texas
  - The Crofoot Research Center, Inc. ( Site 0118), Houston, Texas
- Chile (3):
  - Clinica Arauco Salud ( Site 0200), Santiago, RM
  - Biomedica Research Group ( Site 0202), Santiago
  - Hospital Dr. Hernan Henriquez Aravena ( Site 0203), Temuco
- France (8):
  - Hopital Avicenne ( Site 2302), Bobigny
  - Hopital Saint-Andre ( Site 2307), Bordeaux
  - CHU Hotel Dieu ( Site 2308), Nantes
  - CHU de Nice Hopital Archet 1 ( Site 2303), Nice
  - Hopital Bichat - Claude Bernard ( Site 2309), Paris
  - Hopital Pitie Salpetriere ( Site 2305), Paris
  - Hopital Saint Louis ( Site 2306), Paris
  - Centre Hospitalier de Tourcoing ( Site 2301), Tourcoing
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust ( Site 2105), Brighton, East Sussex
  - Chelsea and Westminster Hospital ( Site 2101), London
  - Royal London Hospital ( Site 2103), London
  - The Royal Free London NHS Foundation Trust ( Site 2102), London
  - North Manchester General Hospital ( Site 2104), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Molina JM, Yazdanpanah Y, Afani Saud A, Bettacchi C, Chahin Anania C, Klopfer SO, Grandhi A, Eves K, Hepler D, Robertson MN, Hwang C, Hanna GJ, Correll T. Brief Report: Efficacy and Safety of Oral Islatravir Once Daily in Combination With Doravirine Through 96 Weeks for Treatment-Naive Adults With HIV-1 Infection Receiving Initial Treatment With Islatravir, Doravirine, and Lamivudine. J Acquir Immune Defic Syndr. 2022 Sep 1;91(1):68-72. doi: 10.1097/QAI.0000000000002879. Epub 2021 Dec 8. PMID 35972855
- [Derived] Molina JM, Yazdanpanah Y, Afani Saud A, Bettacchi C, Chahin Anania C, DeJesus E, Olsen Klopfer S, Grandhi A, Eves K, Robertson MN, Correll T, Hwang C, Hanna GJ, Sklar P. Islatravir in combination with doravirine for treatment-naive adults with HIV-1 infection receiving initial treatment with islatravir, doravirine, and lamivudine: a phase 2b, randomised, double-blind, dose-ranging trial. Lancet HIV. 2021 Jun;8(6):e324-e333. doi: 10.1016/S2352-3018(21)00021-7. Epub 2021 May 14. PMID 34000227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment-naïve participants ≥18 years of age with human immunodeficiency virus type 1 (HIV-1) were enrolled in this study.
Groups:
- Islatravir 0.25 mg: In Part 1, participants were treated once daily (QD) with 0.25 mg islatravir, 100 mg doravirine (DOR), 300 mg lamivudine (3TC), and placebo to doravirine/lamivudine/tenofovir disoproxil fumarate (DOR/3TC/TDF) for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no Protocol-defined Virologic Failure (PDVF) discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 0.25 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144. In Part 4, beginning with Week 144, participants received the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label and continued treatment until Week 192.
- Islatravir 0.75 mg: In Part 1, participants were treated QD with 0.75 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 0.75 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144. In Part 4, beginning with Week 144, participants received the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label and continued treatment until Week 192.
- Islatravir 2.25 mg: In Part 1, participants were treated QD with 2.25 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 2.25 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144. In Part 4, beginning with Week 144, participants received the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label and continued treatment until Week 192.
- DOR/3TC/TDF: In Part 1, participants were treated QD with placebo to islatravir, placebo to DOR, placebo to 3TC, and a fixed dose combination of DOR/3TC/TDF consisting of 100 mg DOR + 300 mg 3TC + 300 mg TDF for a minimum of 24 weeks. In Parts 2 and 3, after a minimum of 24 weeks of treatment, placebo treatments were discontinued and participants received only DOR/3TC/TDF QD open label up to Week 144. In Part 4, beginning with Week 144, participants received the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label and continued treatment until Week 192.
Period: Overall Study
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Started | 31 | 30 | 31 | 31
Treated | 29 | 30 | 31 | 31
Completed | 20 | 24 | 19 | 24
Not Completed | 11 | 6 | 12 | 7
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 5 | 1
Not completed — Physician Decision | 4 | 2 | 5 | 4
Not completed — Screen Failure | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Islatravir 0.25 mg; Islatravir 0.75 mg: In Part 1, participants were treated QD with 0.75 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 0.75 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144. In Part 4, beginning with Week 144, participants received the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label and continued treatment until Week 192.
- Total: Total of all reporting groups
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF | Total
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (13.3) | 30.0 (9.0) | 32.4 (11.8) | 29.4 (8.9) | 31.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 3 | 10
  Male | 30 | 27 | 28 | 28 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 19 | 12 | 15 | 60
  Not Hispanic or Latino | 16 | 11 | 18 | 15 | 60
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 8 | 5 | 25
  White | 24 | 24 | 21 | 24 | 93
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
CD4+ T-Cell Count [Mean (Standard Deviation); unit: cells/mm^3] — Population: Two untreated participants from the Islatravir 0.25 mg treatment group were not analyzed.
  cells/mm^3
    number analyzed (Participants) | 29 | 30 | 31 | 31 | 121
    (all) | 450.8 (170.0) | 538.5 (165.5) | 469.6 (203.3) | 508.5 (206.8) | 492.1 (188.5)
Participants with <=100,000 copies/mL of HIV-1 RNA [Count of Participants; unit: Participants] — Number of participants at screening with <=100,000 copies/mL of HIV-1 RNA
  Participants | 24 | 23 | 23 | 24 | 94
Participants with >100,000 copies/mL of HIV-1 RNA [Count of Participants; unit: Participants] — Number of participants at screening with >100,000 copies/mL of HIV-1 RNA
  Participants | 7 | 7 | 8 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 24
Description: Blood samples were collected and plasma human immunodeficiency virus 1 (HIV-1) ribonucleic acid (RNA) were quantified using a real time polymerase chain reaction (PCR) assay with a lower limit of detection of 40 copies/mL. Missing values were counted as failure.
Time Frame: Week 24
Population: All randomized participants who received at least 1 dose of study treatment and have baseline data for those analyses that require baseline data.
Measure: Number; unit: Percentage of participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
Percentage of participants | 93.1 | 100.0 | 90.3 | 90.3
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — The 95% confidence intervals (CIs) were calculated using stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum (screening HIV-1 RNA ≤100,000 or >100,000 copies/mL); Treatment Difference = 2.9, 95% CI 2-sided [-12.5 to 18.3] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — The 95% CIs were calculated using stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum (screening HIV-1 RNA ≤100,000 or >100,000 copies/mL); Treatment Difference = 9.6, 95% CI 2-sided [-3.8 to 23.0] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = 0.2, 95% CI 2-sided [-16.0 to 16.3] — Islatravir minus DOR/3TC/TDF

2. Primary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48
Description: Blood samples were collected and plasma HIV-1 RNA were quantified using a real time PCR assay with a lower limit of detection of 40 copies/mL. Missing values were counted as failure.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
Percentage of participants | 89.7 | 90.0 | 77.4 | 83.9
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = 6.1, 95% CI 2-sided [-12.2 to 24.4] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = 6.2, 95% CI 2-sided [-12.2 to 24.6] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = -6.1, 95% CI 2-sided [-27.1 to 14.8] — Islatravir minus DOR/3TC/TDF

3. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) up to Week 144
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Time Frame: Up to 144 weeks
Population: All randomized participants who received at least 1 dose of study treatment, corresponding to the study treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
Participants | 26 | 27 | 24 | 27
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 2.6, 95% CI 2-sided [-15.7 to 20.5] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 2.9, 95% CI 2-sided [-15.0 to 20.8] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = -9.7, 95% CI 2-sided [-29.4 to 10.1] — Islatravir minus DOR/3TC/TDF

4. Primary Outcome: Number of Participants Discontinuing Study Drug Due to AEs up to Week 144
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Time Frame: Up to 144 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
Participants | 1 | 0 | 2 | 1
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 0.2, 95% CI 2-sided [-13.4 to 14.5] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = -3.2, 95% CI 2-sided [-16.4 to 8.5] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 3.2, 95% CI 2-sided [-10.8 to 18.1] — Islatravir minus DOR/3TC/TDF

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL up to 24 Weeks After 3TC and Placebo Are Discontinued From the Regimen
Description: Blood samples were collected and plasma HIV-1 RNA were quantified using a real time PCR assay with a lower limit of detection of 40 copies/mL, and missing values were counted as failure. 3TC and placebo are discontinued from the regimen from Week 24 up to Week 52.
Time Frame: Up to 24 weeks after 3TC and Placebo are discontinued from the regimen (up to approximately 60 weeks after initiating treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 27 | 28
Percentage of participants | 86.2 | 90.0 | 88.9 | 96.4
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = -9.7, 95% CI 2-sided [-26.1 to 6.6] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = -6.2, 95% CI 2-sided [-21.5 to 9.1] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = -7.5, 95% CI 2-sided [-23.9 to 8.8] — Islatravir minus DOR/3TC/TDF

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL up to 48 Weeks After 3TC and Placebo Are Discontinued From the Regimen
Description: as for outcome 5
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 27 | 28
Percentage of participants | 62.1 | 56.7 | 59.3 | 60.7
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = 2.2, 95% CI 2-sided [-23.4 to 27.7] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = -3.7, 95% CI 2-sided [-29.6 to 22.1] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in percent response; Test type: Other — [test comment as in outcome 1, analysis 2]; Treatment Difference = -1.3, 95% CI 2-sided [-27.7 to 25.2] — Islatravir minus DOR/3TC/TDF

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL up to 48 Weeks After Starting Open-label Doravirine/Islatravir Regimen (Part 4)
Description: Blood samples were collected and plasma HIV-1 RNA were quantified using a real time PCR assay with a lower limit of detection of 40 copies/mL. Missing values were counted as failure. The percentage of participants with HIV-1 RNA <50 copies in Part 4 are reported.
Time Frame: Up to Week 192
Population: Per protocol, all randomized participants who entered Part 4 and either continued treatment with DOR/ISL from Part 3 or switched from DOR/3TC/TDF in Part 3 to DOR/ISL in Part 4; and received at least 1 dose of study treatment and have baseline data for those analyses that require baseline data were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- DOR/ISL Continued (Part 4): In Part 4, beginning with week 144, participants who received the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label in Part 3 and continued treatment through Week 192.
- DOR/ISL Switch (Part 4): In Part 4, beginning with week 144, participants who received DOR/3TC/TDF QD open label up to Week 144 were switched to the fixed dose combination of doravirine (100 mg)/islatravir (0.75 mg) QD open label and continued treatment until Week 192.
Arm/Group | DOR/ISL Continued (Part 4) | DOR/ISL Switch (Part 4)
Number analyzed (Participants) | 67 | 22
Percentage of participants | 85.1 | 95.5

8. Secondary Outcome: Change From Baseline in Mature T-helper (CD4+ T)-Cell Count at Week 24
Description: Blood samples were collected and cluster of differentiation (CD4)+ T-cell counts were performed, where baseline measurements are defined as the Day 1 value, and baseline values were carried forward for participants who discontinue due to lack of efficacy. Post-baseline data were collected after the first dose of study medication through 14 days after the last dose of study medication.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
cells/mm^3 | 220.5 [170.3 to 270.8] | 192.8 [117.9 to 267.7] | 142.9 [89.9 to 196.0] | 142.1 [105.7 to 178.5]
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = 78.4, 95% CI 2-sided [18.8 to 138.1] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = 50.7, 95% CI 2-sided [-31.7 to 133.1] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = 0.8, 95% CI 2-sided [-63.0 to 64.7] — Islatravir minus DOR/3TC/TDF

9. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 48
Description: Blood samples were collected and CD4+ T-cell counts were performed, where baseline measurements are defined as the Day 1 value, and baseline values were carried forward for participants who discontinue due to lack of efficacy. Post-baseline data were collected after the first dose of study medication through 14 days after the last dose of study medication.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
cells/mm^3 | 182.0 [119.6 to 244.5] | 183.0 [124.7 to 241.2] | 100.7 [25.0 to 176.3] | 181.4 [137.2 to 225.6]
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = 0.6, 95% CI 2-sided [-74.1 to 75.3] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = 1.5, 95% CI 2-sided [-70.7 to 73.8] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -80.8, 95% CI 2-sided [-165.6 to 4.0] — Islatravir minus DOR/3TC/TDF

10. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 96
Description: as for outcome 9
Time Frame: Baseline and Week 96
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
cells/mm^3 | 243.4 [165.5 to 321.3] | 161.3 [90.2 to 232.4] | 136.5 [57.0 to 216.0] | 268.9 [188.5 to 349.3]
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -25.5, 95% CI 2-sided [-134.8 to 83.8] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -107.6, 95% CI 2-sided [-212.1 to -3.1] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -132.4, 95% CI 2-sided [-242.9 to -21.9] — Islatravir minus DOR/3TC/TDF

11. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 144
Description: as for outcome 9
Time Frame: Baseline and Week 144
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 31 | 31
cells/mm^3 | 204.4 [102.0 to 306.7] | 209.0 [111.5 to 306.6] | 162.9 [70.2 to 255.5] | 270.0 [183.2 to 356.8]
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -65.6, 95% CI 2-sided [-195.3 to 64.0] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -61.0, 95% CI 2-sided [-188.7 to 66.8] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Treatment difference in T-cell count; Test type: Other — The 95% CI for mean difference in CD4 change was based on t-distribution; Treatment Difference = -107.1, 95% CI 2-sided [-231.2 to 16.9] — Islatravir minus DOR/3TC/TDF

12. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 192 (Part 4)
Description: Blood samples were collected and CD4+ T-cell counts were performed, where baseline measurements are defined as the Week 144 value. The change from baseline in CD4+ T-cell count at Week 192 (Part 4) are reported.
Time Frame: Baseline and Week 192
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | DOR/ISL Continued (Part 4) | DOR/ISL Switch (Part 4)
Number analyzed (Participants) | 57 | 21
cells/mm^3 | 3.8 [-1.9 to 9.5] | -3.4 [-12.0 to 5.2]

13. Secondary Outcome: Number of Participants Experiencing AEs Through 24 Weeks After 3TC and Placebo Are Discontinued From the Regimen
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. 3TC and placebo are discontinued from the regimen from Week 24 up to Week 52.
Time Frame: Up to 24 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 27 | 28
Participants | 18 | 20 | 14 | 16
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 4.9, 95% CI 2-sided [-20.3 to 29.6] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 9.5, 95% CI 2-sided [-15.4 to 33.5] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = -5.3, 95% CI 2-sided [-30.6 to 20.7] — Islatravir minus DOR/3TC/TDF

14. Secondary Outcome: Number of Participants Discontinuing Study Drug Due to AEs Through 24 Weeks After 3TC and Placebo Are Discontinued From the Regimen
Description: as for outcome 13
Time Frame: Up to 24 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF
Number analyzed (Participants) | 29 | 30 | 27 | 28
Participants | 0 | 0 | 2 | 1
Statistical Analysis 1: Comparison: Islatravir 0.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = -3.6, 95% CI 2-sided [-17.9 to 8.5] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 2: Comparison: Islatravir 0.75 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = -3.6, 95% CI 2-sided [-17.9 to 8.2] — Islatravir minus DOR/3TC/TDF
Statistical Analysis 3: Comparison: Islatravir 2.25 mg vs DOR/3TC/TDF; Difference in % Islatravir vs DOR/3TC/TDF; Test type: Other — Based on Miettinen & Nurminen method; Difference in % = 3.8, 95% CI 2-sided [-11.5 to 20.6] — Islatravir minus DOR/3TC/TDF

15. Secondary Outcome: Number of Participants Experiencing AEs From Week 96 Through Study Duration
Description: as for outcome 4
Time Frame: Week 96 up to Week 192
Population: Per protocol, all randomized participants who received at least 1 dose of open label study treatment in Part 3 or Part 4, corresponding to the study treatment they actually received were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Islatravir 0.25 mg; Islatravir 0.75 mg: In Part 1, participants were treated QD with 0.75 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 0.75 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144.
- Islatravir 2.25 mg: In Part 1, participants were treated QD with 2.25 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 2.25 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144.
- DOR/3TC/TDF: In Part 1, participants were treated QD with placebo to islatravir, placebo to DOR, placebo to 3TC, and a fixed dose combination of DOR/3TC/TDF consisting of 100 mg DOR + 300 mg 3TC + 300 mg TDF for a minimum of 24 weeks. In Parts 2 and 3, after a minimum of 24 weeks of treatment, placebo treatments were discontinued and participants received only DOR/3TC/TDF QD open label up to Week 144.
- DOR/ISL Continued: In Part 4, beginning with week 144, participants who received the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label in Part 3 and continued treatment through Week 192.
- DOR/ISL Switch: In Part 4, beginning with week 144, participants who received DOR/3TC/TDF QD open label up to Week 144 were switched to the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label and continued treatment until Week 192.
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF | DOR/ISL Continued | DOR/ISL Switch
Number analyzed (Participants) | 29 | 30 | 31 | 31 | 67 | 22
Participants | 12 | 19 | 11 | 12 | 36 | 14

16. Secondary Outcome: Number of Participants Discontinuing Study Drug Due to AEs From Week 96 Through Study Duration
Description: as for outcome 4
Time Frame: Week 96 up to Week 192
Population: Per protocol, all randomized participants who received at least 1 dose of open label study treatment in Part 3 or Part 4, corresponding to the study treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 0.25 mg | Islatravir 0.75 mg | Islatravir 2.25 mg | DOR/3TC/TDF | DOR/ISL Continued | DOR/ISL Switch
Number analyzed (Participants) | 29 | 30 | 31 | 31 | 67 | 22
Participants | 1 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants Experiencing AEs During Open Label Doravirine/Islatravir Treatment After Week 144 up to Week 192 (Part 4)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experienced AEs during Part 4 are reported.
Time Frame: Week 144 up to Week 192
Population: Per protocol, all randomized participants who entered Part 4 and either continued treatment with DOR/ISL from Part 3 or switched from DOR/3TC/TDF in Part 3 to DOR/ISL in Part 4; and received at least 1 dose of study treatment, corresponding to the study treatment they actually received were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- DOR/ISL Continued (Part 4): In Part 4, beginning with week 144, participants who received the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label in Part 3 and continued treatment through Week 192.
- DOR/ISL Switch (Part 4): In Part 4, beginning with week 144, participants who received DOR/3TC/TDF QD open label up to Week 144 were switched to the fixed dose combination of doravirine (100mg)/islatravir (0.75mg) QD open label and continued treatment until Week 192.
Arm/Group | DOR/ISL Continued (Part 4) | DOR/ISL Switch (Part 4)
Number analyzed (Participants) | 67 | 22
Participants | 36 | 14

18. Secondary Outcome: Number of Participants Discontinuing Study Drug Due to AEs During Open Label Doravirine/Islatravir Treatment After Week 144 up to Week 192 (Part 4)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who discontinued the study drug due to AEs in Part 4 are reported.
Time Frame: Week 144 up to Week 192
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL Continued (Part 4) | DOR/ISL Switch (Part 4)
Number analyzed (Participants) | 67 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: For All-Cause Mortality: from randomization up to 198 weeks. For AEs: from first treatment up to 198 weeks.
Description: The population analyzed for All-Cause Mortality was all randomized participants. The population analyzed for AEs was all randomized participants who received at least 1 dose of study treatment, corresponding to the study treatment they actually received.
Groups:
- Islatravir 0.25mg; Islatravir 0.75mg: In Part 1, participants were treated QD with 0.75 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 0.75 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144.
- Islatravir 2.25mg: In Part 1, participants were treated QD with 2.25 mg islatravir, 100 mg DOR, 300 mg 3TC, and placebo to DOR/3TC/TDF for a minimum of 24 weeks. In part 2, after receiving at least 24 weeks of study intervention, participants with HIV-1 RNA <50 copies/mL and no PDVF discontinued treatment of 3TC and placebo to DOR/3TC/TDF. Part 2 assessed ISL 2.25 mg (blind maintained) + DOR QD. After all participants had received at least 48 weeks of study intervention and the islatravir dose was selected, all participants in the islatravir group were switched to the selected dose 0.75 mg (between week 60 and week 84). Part 3 assessed Islatravir 0.75 mg + DOR QD open label through Week 144.
Arm/Group | Islatravir 0.25mg | Islatravir 0.75mg | Islatravir 2.25mg | DOR/3TC/TDF | DOR/ISL Continued | DOR/ISL Switch
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 1/31 | 0/67 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/29 | 6/30 | 2/31 | 4/31 | 2/67 | 1/22
Other Adverse Events (participants affected / at risk) | 22/29 | 26/30 | 23/31 | 22/31 | 21/67 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islatravir 0.25mg (N=29) | Islatravir 0.75mg (N=30) | Islatravir 2.25mg (N=31) | DOR/3TC/TDF (N=31) | DOR/ISL Continued (N=67) | DOR/ISL Switch (N=22)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Long QT syndrome congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islatravir 0.25mg (N=29) | Islatravir 0.75mg (N=30) | Islatravir 2.25mg (N=31) | DOR/3TC/TDF (N=31) | DOR/ISL Continued (N=67) | DOR/ISL Switch (N=22)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (8) | 3 (3) | 8 (11) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (6) | 3 (3) | 3 (5) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (5) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 7 (7) | 1 (1) | 5 (7) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (4) | 9 (10) | 2 (2) | 7 (14) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 2 (2) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Syphilis (Infections and infestations) | 6 (6) | 8 (8) | 2 (2) | 6 (7) | 4 (4) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (4) | 3 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (4) | 3 (5) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (4) | 4 (4) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (5) | 5 (6) | 4 (5) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03272347/Prot_SAP_000.pdf